CLINICAL TRIAL: NCT03124693
Title: Accuracy of Noninvasive Hemoglobin Measurement (SpHb) Using Rainbow DCI Pulse Oximeter Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR-17412-TORP0001
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Healthy; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Group (Experimental): All subjects are enrolled into the test group and all subjects received the Rainbow DCI pulse oximeter sensor.
  Interventions: Device: Rainbow DCI pulse oximeter sensor

INTERVENTIONS:
Device: Rainbow DCI pulse oximeter sensor

SUMMARY:
In this study, the concentration of hemoglobin within the subject's blood is affected by fluid status changes. The fluid status is affected by fluid loss during surgery for hospitalized study subjects or controlled administration of fluids intravenously for healthy study volunteers. The accuracy of a noninvasive hemoglobin sensor(s) will be assessed by comparing with blood sample analysis.

ELIGIBILITY:
Healthy Volunteers

Inclusion Criteria:

* Has physical status between ASA 1 or 2
* Able to communicate in English

Exclusion Criteria:

* Pregnant or sexually active without birth control.
* Hemoglobin less than 11g/dL
* Known alcohol or drug abuse
* Skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection
* Nail polish
* Head injury with loss of consciousness within the last year
* Known neurological and psychiatric conditions.
* Known concurrent chronic usage of psychoactive or anti-convulsive drugs within the last 90 days, or use in the last 7 days (i.e. tricyclic antidepressants, MAO inhibitors, lithium, neuroleptics, anxiolytics or antipsychotics. Except SSRIs
* Subject has any medical condition which, in the judgement of the investigator, renders them inappropriate for participation in this study, such as Reynauds syndrome
* Hypertension: Systolic BP >= 140 mmHg or Diastolic BP >= 90 mmHg
* Baseline heart rate <50 beats per minute

Surgical Subjects

Inclusion Criteria:

* Age > 18 years old
* Scheduled for surgery requiring frequent schedule blood draws as a part of their routine care

Exclusion Criteria:

* Pregnant or lactating women
* Skin abnormalities at the planed application sites that would interfere with transilluminating the finger, or other measurement sites, like burns, scar tissue, nail polish, infections etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-08-12 (Actual); Primary Completion 2008-09-09 (Actual); Study Completion 2008-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Masimo Clinical Lab, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Mayo Clinic, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: All subjects are enrolled into the test group and all subjects received the Rainbow DCI pulse oximeter sensor.
  Rainbow DCI pulse oximeter sensor
Period: Overall Study
Arm/Group | Test Group
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square (Arms) error value.
Time Frame: Up to 24 hours
Measure: Number; unit: g/dL
Arm/Group | Test Group
Number analyzed (Participants) | 90
g/dL | 0.9

ADVERSE EVENTS:
Arm/Group | Test Group
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less